CLINICAL TRIAL: NCT07116616
Title: A Phase 1/2, Open-label, Multicenter Study of mRNA-2808 in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of mRNA-2808 in Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-2808-P101
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: relapsed or refractory multiple myeloma; RRMM; multiple myeloma; MM
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-2808 (Experimental): Participants will receive mRNA-2808.
  Interventions: Drug: mRNA-2808

INTERVENTIONS:
Drug: mRNA-2808 — intravenous

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of mRNA-2808 in participants with relapsed or refractory multiple myeloma (RRMM).

ELIGIBILITY:
Key Inclusion Criteria:

* RRMM with prior exposure to a proteasome inhibitor, an immunomodulatory drug (IMiD), and an anti-cluster of differentiation (CD38) monoclonal antibody.
* Measurable disease defined as at least 1 of the following:

  * Serum M-protein ≥0.5 grams/deciliter
  * Urine M-protein ≥200 milligrams (mg)/24-hour
  * Involved free light chain (FLC) ≥100 mg/liter and an abnormal FLC ratio
  * Plasmacytoma with a single diameter ≥2 centimeters
  * Bone marrow plasma cells >30%

Key Exclusion Criteria:

* Known central nervous system (CNS) myeloma or clinical signs and symptoms of CNS involvement of myeloma.
* Active plasma cell leukemia, defined as peripheral blood plasma cells ≥20%.
* Radiotherapy or cytotoxic chemotherapy within 2 weeks prior to Day 1 (Baseline), except palliative radiotherapy of limited field is permissible within 2 weeks after discussion with the Sponsor medical monitor.
* Antibody-based immunotherapy (monoclonal antibody, bispecific antibody, antibody drug conjugate) within 21 days prior to Day 1 (Baseline).
* Proteasome inhibitor therapy or immunomodulatory agent within 14 days prior to Day 1 (Baseline).
* Autologous hematopoietic cell transplant within 100 days prior to Day 1 (Baseline).
* Allogeneic hematopoietic cell transplant within 180 days prior to Day 1 (Baseline).
* Genetically modified adoptive autologous or allogeneic cellular therapy (for example, chimeric antigen receptor T cell, chimeric antigen receptor natural killer) within 12 weeks prior to Day 1 (Baseline).
* Corticosteroid therapy ≥140 mg prednisone or equivalent cumulative dose within 14 days prior to Day 1 (Baseline).

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2030-06-17 (Estimated); Study Completion 2032-06-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicity | Up to 28 days
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 15 months

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 1 year
Area Under the Concentration-time Curve (AUC) | Up to 1 year
Maximum Effect/Concentration of the Expressed Protein (Emax) | Up to 1 year
Area Under the Effect Concentration (AUEC) | Up to 1 year
Overall Response Rate (ORR) | Up to 3 years
Duration of Response (DOR) | Up to 3 years
Progression-free Survival (PFS) based on International Myeloma Working Group (IMWG) Response Criteria | Up to 3 years
Overall Survival (OS) | Up to 3 years
Number of Participants with Minimal Residual Disease Negativity Status | Up to 3 years
Number of Participants with Antibodies to mRNA-2808 Derived Proteins | Up to 1 year
Number of Participants with Antibodies to mRNA-2808 Components | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - UCSF, San Francisco, California
  - Emory University Hospital, Atlanta, Georgia
  - Mass General Brigham, Boston, Massachusetts
  - Tisch Cancer Institute at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Penn Medicine, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The Medical College of Wisconsin, Milwaukee, Wisconsin